CLINICAL TRIAL: NCT00194636
Title: Effectiveness 0f Sympathetic Plexus Block on Male Pelvic Pain (Prostatitis, Prostatodynia)
Brief Title: Effectiveness of Sympathetic Plexus Block on Male Pelvic Pain (Prostatitis, Prostatodynia)
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: PI health issues
Sponsor: University of Washington (Other)
Collaborators: Paul G. Allen Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24993
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2007-10

CONDITIONS: Chronic Male Pelvic Pain Syndrome; Prostatitis
Keywords: Prostatitis; Chronic Male Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis | interventions — Nerve Block

INTERVENTIONS:
Procedure: nerve block

SUMMARY:
The purpose of this study is to investigate, by means of a temporary sympathetic nerve block, the involvement of the sympathetic nervous system in Chronic Pelvic Pain Syndrome (CPPS). This study may also result in a new therapeutic approach for male CPPS.

DETAILED DESCRIPTION:
Male pelvic pain is a common urological complaint. Oftentimes patients are given the diagnosis of chronic prostatitis. Although the term "chronic prostatitis" is commonly associated with infection, less than 5% of men presenting with pelvic pain are found to have evidence of urogenital infection with common pathogens. Because no etiology can usually be associated with the pain, chronic idiopathic prostatitis is now called male chronic pelvic pain syndrome (CPPS). Options proposed for the treatment of male CPPS have had limited and variable success rates.

Although several abnormalities of the nervous system have been proposed as possible causes of CPPS, the clinical nature of the disease suggests involvement of the sympathetic nervous system. The sympathetic nervous system may be involved in many regional pain syndromes, and in such situations, the term "sympathetically maintained pain" has been used with complex regional pain syndromes. Block of the sympathetic nerves supplying this region is commonly used to detect sympathetic nervous system involvement.

Sympathetic nerve blocks have been used in some clinical studies involving pelvic pain but most of these studies included cancer patients with pelvic pain. The type of sympathetic blocks used for pelvic pain is superior hypogastric plexus block and it involves instillation of neural blocking agents such as local anesthetic agents in the region of the plexus, usually under fluoroscopic control. Nociceptive afferent transmission from pelvic viscera is probably via the superior hypogastric plexus. This treatment option has not been systematically used for male CPPS.

In this study, a temporary block of the superior hypogastric plexus with bupivacaine will be used to assess the degree of sympathetic block with some electrodiagnostic tests. After the temporary nerve block, the analgesic efficacy will be monitored. Therefore, in this study, we hope not only to explain the sympathetic nature of the disease in more concrete terms but also propose a new therapeutic approach for male CPPS.

Men with a diagnosis of non-bacterial chronic pelvic pain who have not responded to treatment will be asked to participate in this study. The subjects will be randomly assigned to receive either active medication as the sympathetic plexus block or placebo. All other study elements will be identical for both groups.

Visit 1 will take approximately 4 hours at the University of Washington Medical Center Urology Clinic.

* First, the study will be explained in detail to the subject. Any questions he has will be answered and he will be given the study consent to read and sign.
* Next, the subject will be asked to fill out baseline questionnaires. They are Demographic Questionnaire, Baseline Symptom Questionnaire, NIH Symptom Index-Baseline, AUA Symptom Score, short version of the Perceived Stress Scale (PSS) and Pain Drawing. A sexual function questionnaire, the International Index of Erectile Function (IIEF) will also be administered. After completing the questionnaires, the subject will have a physical and neurological exam.
* Blood draw: An 20 gauge needle will be inserted to antecubital vein and fixed with tape. The subject will lie down on the examination table for 20 minutes and then have approximately 10 cc of blood drawn, via the needle, to be used for baseline plasma catecholamine, corticosteroid and acetylcholine levels. Plasma catecholamine measurement is a biochemical parameter to evaluate sympathetic nervous system. Corticosteroids are stress-related hormones and acetylcholine is an important neurotransmitter related to autonomic nervous system.
* We will next ask the patient to stand. After he has been standing for 5 minutes, another 10cc of blood will be drawn then the needle removed. This blood will be used to measure the same hormonal parameters, as above, but after the nervous system has been activated by standing.
* Prostate massage and rectal/prostate exam: The subject will undergo a rectal and prostate examination with massage of the prostate and expressions of prostatic fluids. The subject will be asked to come with a full bladder and asked to urinate about 5 cc into a small container. He will then be asked to urinate 20 cc into a second container and save the rest in his bladder. The subject will then undergo a rectal examination and prostate massage and if possible obtaining expressed prostatic secretions from the tip of the penis. The subject will then be asked to urinate a third time approximately 10 cc into a sterile container. Specimens will be used for microbiologic and biochemical studies.
* Semen analysis: We will ask the subject to provide a semen sample through masturbation. A private room, with a lockable door, will be provided for this purpose.
* Some of the specimens collected at this visit will be saved for future use for possible biochemical studies. These studies will be available only to the investigators involved in this study and given to no one else. If in the future, it is deemed by the investigators to be scientifically and clinically valuable, these specimens may be used for genetic testing for genes that make one susceptible to pelvic pain syndromes such as prostatitis. If genetic testing is ever considered in the future, the subject will be contacted and asked to sign another consent form. The consent will state the exact nature of the testing and clearly explain why it is being done.
* Electrodiagnostic tests: These are the tests to evaluate the sympathetic nervous system tone and also sensations in several parts of the body including the genital area. The first electrodiagnostic test will involve a battery controlled instrument called Episcan. It measures the skin conductivity response on several sites of the body. We will apply this test on penis, scrotum, genital area, perineum, hands and feet. It is a painless and non-invasive test and it does not require any stimulation.
* The second part of the electrodiagnostic tests will involve use of another battery controlled instrument called Neurometer. This is a painless procedure that detects and localizes abnormalities of sensation in several body parts. We will apply this test on both feet, hands, penis, scrotum, genital area and perineum. Three different types of stimuli with different frequencies will be delivered to determine the sensory threshold in each of these areas tested.
* The third test will be the measurement of temperature sensations in the painful area, the perineum and left hand. In order to measure temperature sensation, a small probe capable of changing temperature will be placed on these areas. The ability to discriminate temperature changes will be determined as well as the subjective discomfort produced by the temperature changes. A computer assisted device called Thermal Sensory Analyzer will be used for that purpose.
* Then, the subject will have sympathetic skin response and evoked cavernous activity measurements. These tests reflect the state of the sympathetic nervous system in the evaluated body part. The subject will be in the supine position throughout. Two 28 ga. concentric needle electrodes will be placed into the side of the penis. Six surface electrodes will be placed on the penile skin, on scrotum, on perineum and on abdominal skin as recording electrodes. Eight other surface electrodes will be placed on the back and inner sides of both feet and both hands. After the electrodes are placed, spontaneous electrical activity will be recorded for 5 minutes. After obtaining spontaneous surface and needle electrode recordings, the right wrist (median nerve) will be stimulated a small amount of current. Median nerve stimulation is a routine method used to stimulate the nervous system in order to record electrical skin responses. After the stimulation of the median nerve, evoked responses will be acquired through the existing electrodes. The stimulus to the median nerve will be repeated.
* After this test, all the electrodes will be taken out and two needle electrodes as used in the penis will be inserted into the cremasteric muscles on both sides. These are the muscles surrounding the vessels that supply testicles. Then, inner side of right thigh will be stimulated a small amount of current to evoke cremasteric muscle reflexes. This reflex shows the state of sympathetic nerves that supply testicles and scrotum. These tests will be useful to assess the degree of sympathetic nerve blockage by comparing to the tests after the instillation.
* At the end of the visit, the subject will be given a voiding diary and plastic urinal. We will ask him to measure and record his urine output for any 3 consecutive days during the coming week.

VISIT 2 will take approximately 4 hours at the University of Washington Medical Center Urology Clinic.

* In this visit, the subject will be taken into fluoroscopy unit in the Urology clinic. The subject will lie in the prone position and will receive a subcutaneous injection of 1% lidocaine without epinephrine.
* Then, under radiologic guidance, two needles (22-G Chiba) will be placed via a bilateral posterior approach such that the tips of both needles lie anterior to the L5/S1 vertebrae. Placement of the needle will be monitored closely in order to avoid any other anatomical structures. The exact locations of needles will be confirmed with injection of radiopaque solution (Isovue-200) under fluoroscopy. After ensuring correct needle placement, 0.5% levobupivacaine, 10ml will be injected in each needle in the study group and 0.9% NaCl solution, 10ml in the control group. Routine monitoring (ECG/blood pressure, pulse oximetry) will be used throughout the procedure and for 30 minutes after the procedure.
* One hour following the procedure, the blood draw, urine collection (without prostate massage) and the electrodiagnostic tests as in the first visit will be repeated in order to assess the degree of block. The subjects will be given another copy of the voiding diary to fill out during the next week.

VISIT 3 will take about 4 hours and will take place one week following the procedure. The sympathetic blockage will be assessed for its side effects on sexual and voiding function with a through physical and neurological examination. The pain questionnaires NIH SX-Follow/up, AUA-Symptom Score, IIEF, PSS and Pain Drawing and the electrodiagnostic tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Men with Chronic Pelvic Pain Syndrome who, for the past year, have not responded to standard pain treatment modalities.

Exclusion Criteria:

* Urinary tract infection with common pathogens
* Treatment for prostate, bladder, renal, or other urinary malignancies.
* Back pain or rectal pain only
* Psychotic or suicidal men
* Post-surgical pain
* Pain from another source in genital the tract such as kidney stones or neoplasm
* Having had radiation therapy
* History of genitourinary tuberculosis
* Neurological abnormalities such as stroke, brain tumors, spinal tumors, spinal cord injury and Parkinson's or Alzheimer's disease.
* Drug allergies
* Use of any drugs, such as antihypertensives, that would interfere with biochemical and electrodiagnostic tests.
* Bleeding and clotting disorders such as factor deficiencies or anticoagulant drug use.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2006-11

PRIMARY OUTCOMES:
change in symptom score; reflected in NIH-Symptom Index (CPSI) at Block Assessment Visit

SECONDARY OUTCOMES:
AUA score at Block Assessment Visit

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Berger, MD, Principal Investigator — Professor of Urology
Locations (1):
- University of Washington - Urology Clinic, Seattle, Washington, United States